CLINICAL TRIAL: NCT03487718
Title: Ridge Preservation With Leukocyte Platelet Rich Fibrin: A Clinical, Radiographic, and Histomorphometric Study.
Brief Title: A 14 Weeks Longitudinal Study to Investigate the Effect of Leukocyte- Platelet Rich Fibrin Plug on the Quality of the Newly Formed Bone in Ridge Preservation Procedure Following a Tooth Extraction. It is a Clinical, Radiographic and Histomorphometric Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firas Al Yafi (Other)
Responsible Party: Sponsor-Investigator, Firas Al Yafi, Periodontology Resident, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0815-F2L
Record Dates: First submitted 2018-03-14; First posted 2018-04-04 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Alveolar Ridge Preservation; Tooth Extraction
Keywords: Platelet-Rich Fibrin; high-density polytetrafluoroethylene membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control group (Active Comparator): Under the effect of local anesthetic tooth will be extracted then a d-PTFE membrane will be used to cover the socket without any bone graft material to preserve the ridge.
  Interventions: Device: d-PTFE membrane
- Test group (Experimental): Under the effect of local anesthetic tooth extraction will be followed by the collection of about 50 ml of the patient's venous blood, then without adding any anticougulant the blood will be spun to make a plug. The Leukocyte platelet rich fibrin plug + d-PTFE membrane will be used to preserve the ridge.
  Interventions: Biological: Leukocyte platelet rich fibrin plug + d-PTFE membrane

INTERVENTIONS:
Biological: Leukocyte platelet rich fibrin plug + d-PTFE membrane — Following tooth extraction, an autologous leukocyte platelet rich fibrin plug will be placed in the socket and covered with a d-PTFE membrane
  Arms: Test group
Device: d-PTFE membrane — Following tooth extraction, the socket will be covered with a d-PTFE membrane
  Other Names: Cytoplast
  Arms: Control group

SUMMARY:
This 14 weeks longitudinal study will be conducted from March 2018 to June 2020, with a 40 participants. No subjects has received placebo medication at any point in the research procedures.

Null hypothesis: The use of L-PRF plug, in combination with non-resorbable, open barrier membrane technique to fill the extraction sockets will have no effect on the quality of the newly formed bone nor on the dimensional changes of the ridge, compared to non-resorbable, open barrier membrane technique with natural blood clot.

DETAILED DESCRIPTION:
This 14 weeks longitudinal study was conducted from March 2018 to June 2020, with a 27 participants. No subjects has received placebo medication at any point in the research procedures.

The proposed sample population has been recruited from the patient population of the University of Kentucky College of Dentistry clinics and the patient must have had an unsalvageable tooth that was planned for extraction and delayed implant placement and was assigned into a control group and a test group by chance. Fifteen extraction socket sites of the test group were filled with autogenous L-PRF Plug (Intralock) and d-PTFE membrane (Cytoplast) was laid on the top to seal the extraction socket. In the control group, d-PTFE membrane (Cytoplast) was laid on the top of twelve extraction sockets to allow natural blood clot formation in the extraction socket.

The primary aim is to assess the quality of the newly formed bone at 14 weeks the time of implant placement by comparing the percentage of new vital bone in the histomorphometric analysis. The second aim was to assess the horizontal and vertical changes of the residual bony ridge using Cone Bean Computerized Tomography (CBCT) analysis at baseline immediately after tooth extraction at 12 weeks of healing.

Null hypothesis: The use of L-PRF plug, in combination with non-resorbable, open barrier membrane technique to fill the extraction sockets will have no effect on the quality of the newly formed bone nor on the dimensional changes of the ridge, compared to non-resorbable, open barrier membrane technique with natural blood clot.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have an unsalvageable tooth that is planned for extraction and delayed implant placement.
* The tooth should be free of acute odontogenic infections.
* Extraction sockets with minimal to moderate bony defect.

Exclusion Criteria:

* Any patient who is planned for full mouth extraction.
* Heavy smoker (more than 10 cigarettes a day).
* History of malignancy, chemotherapy, radiation therapy.
* Immunosuppressive disease.
* Uncontrolled systemic disease.
* Any contraindications to surgical procedures.
* Females who are pregnant or breastfeeding.
* For multi-rooted teeth, if the most coronal part of the interradicular septum is less than 5 mm below the crest of the bone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mhdfiras Al Yafi, DDS, Principal Investigator — University of Kentucky College of Dentistry
Locations (1):
- Univerisity of Kentucky College of Dentistry, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from the University of Kentucky College of Dentistry clinics between Mar 2018 and Dec 2019.
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 12 | 15
Completed | 11 | 11
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Test Group | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 9 | 12 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 13 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Quality of the Newly Formed Bone
Description: Histomorphometric analysis will be performed on a bone core sample harvested at the time of implant placement.
Time Frame: The bone sample was harvested at 14 weeks from the baseline visit (extraction of tooth).
Measure: Mean (Standard Deviation); unit: Percentage of newly formed bone
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 11 | 11
Percentage of newly formed bone | 24.14 (16.26) | 19.12 (10.57)

2. Secondary Outcome: Dimensional Changes of the Alveolar Ridge (Ridge Width)
Description: Two Cone Bean Computerized Tomography (CBCT) measurements were compared to perform the analysis.
Time Frame: The baseline CBCT after tooth extraction and 12 weeks CBCT after extraction.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 11 | 11
mm | 0.81 (0.59) | 1.22 (0.97)

ADVERSE EVENTS:
Time Frame: Adverse event data collection was performed over 14 weeks for each patient, The patient's visits included: • Baseline visit. • Week-one visit. • Week-four visit. • Week-twelve visit. • Week-fourteen visit. All procedures described above were standard of care except for bone core biopsy which was research related.
Description: Subjects were monitored for any adverse reactions throughout the study. All adverse events were managed and documented by the principal investigator.
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-03-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03487718/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03487718/SAP_001.pdf